CLINICAL TRIAL: NCT02748551
Title: Prospective Multicenter Study on Laparoscopic Gastric Cancer Surgery Compared With Open Surgery for Locally Advanced Gastric Cancer
Brief Title: A Comparison Laparoscopic With Open Gastric Cancer Surgery for Locally Advanced Gastric Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Moscow Clinical Scientific Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MKNC 01/2016
Record Dates: First submitted 2016-04-10; First posted 2016-04-22 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; locally advanced gastric cancer; laparoscopic surgery; laparoscopic procedure; comparison laparoscopic with open procedure; multicenter trials
MeSH Terms: conditions — Stomach Neoplasms | interventions — Laparoscopy; Conversion to Open Surgery

ARMS (2):
- Laparoscopic surgery (Experimental): Traditional open procedure for patient with locally advanced gastric cancer
  Interventions: Procedure: Open Surgery
- Open surgery (Active Comparator): Minimum invasive procedure (laparoscopic) for patient with locally advanced gastric cancer
  Interventions: Procedure: Laparoscopic procedures

INTERVENTIONS:
Procedure: Laparoscopic procedures — Laparoscopic surgery
  Arms: Open surgery
Procedure: Open Surgery — Open surgery
  Arms: Laparoscopic surgery

SUMMARY:
Nowadays, the proportion of patients with locally advanced gastric cancer is estimated up to 90 percent of all gastric cancer cases in Russian Federation. Surgical procedure with D2 Lymphadenectomy is the main option for treatment. Conventional open approach is still the current standard for advanced gastric cancer. Laparoscopic procedures for gastric cancer as minimally invasive surgery has gained popularity for the treatment of early gastric cancer in East Asia. Several studies indicated that laparoscopic procedures both total and subtotal gastrectomy with D2 lymphadenectomy is a technically feasible and safe procedure by experienced surgeons in high-volume specialized hospitals. However, lack of solid evidence on the oncologic efficacy.

Starting clinical trials for evaluate safety of oncology laparoscopic subtotal gastrectomy for locally advanced gastric cancer. Aim of this trial is show safety, feasibility and oncologic efficacy of Laparoscopic radical surgical procedures both total and subtotal gastrectomy for treatment gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* ECOG 0-1
* ASA I-III
* Histologically proven cancer of the stomach cT 2-4a(clinical stage tumor), N0-3, M0 at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual Seventh Edition
* Preoperative examination with no distant metastasis, no significantly enlarged lymph nodes around abdominal main artery, and tumor not a direct violation of the pancreas, spleen and other surrounding organs
* The gastric tumors are located in the stomach, are macroscopically resectable by subtotal or total gastrectomy with D2 lymph node dissection.
* Written informed consent

Exclusion Criteria:

* Clinically apparent distant metastasis
* Free cancer cells
* Bulky lymph node metastasis is detected by abdominal CT
* Previous treatment with radiation therapy for any tumors.
* Previous surgery for the present disease
* Pregnancy
* Psychiatric disease

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
"Major" Surgical Morbidity | 21 days.
  "Major" Surgical morbidity is defined as the complication grade on III-V Clavien-Dindo Classification which occurs with-in postoperative 21 days, extension of hospitalization and re-hospitalization. It is necessary to evaluate the complication and if it occurs during the hospitalization, it is required to record complication name, date of on-set (postoperatively), grade on Clavien-Dindo Classification and treatment for complication.

SECONDARY OUTCOMES:
3-year progression-free survival | 36 months
  In terms of locally advanced gastric cancer, to evaluate the progression-free survival rate in laparoscopic gastrectomy with D2 lymph node dissection at postoperative 3 years compared with open procedures
3-year overall survival | 6, 12, 18, 24, 30 and 36 months
  In terms of locally advanced gastric cancer, to evaluate the overall survival rate in laparoscopic gastrectomy with D2 lymph node dissection at postoperative 3 years compared with open procedures
5-year overall survival rate | 6, 12, 18, 24, 30, 36, 48 and 60 months
  In terms of locally advanced gastric cancer, to evaluate the overall survival rate in laparoscopic gastrectomy with D2 lymph node dissection at postoperative 5 years compared with open procedures
Surgical Mortality | 90 days
  It is defined as the death within postoperative 90 days regardless of postoperative reason.
Peri-operative blood loss | 1 day
  Minimally-invasive surgery is associated with less peri-operative blood loss. Blood loss will be measured in milliliters and average blood loss will be compared to the conventional 'open' group.
Postoperative recovery index | 10 days
  Time to first ambulation, flatus, liquid diet, soft diet, and duration of hospital stay are used to assess the postoperative recovery course The amount of abdominal drainage and blood transfusion are also recorded
Pain scores | up to 3 days after surgery
  Pain scores based on a visual analog scale the day of surgery and the subsequent 3 days postoperative 1 days, 2 days, 3 days
Postoperative quality of life | 6, 12, 18, 24, 30 and 36 months
  Both the European Organization for Research and Treatment of Cancer (EORTC) C30 and STO22 are analyzed with quality of life
long-term surgical morbidity | 21days - 36 months after surgery
  Surgical morbidity is defined as the events which occurs with-in postoperative 21 days - 36 months after surgery. It is necessary to evaluate the complication, it is required to record complication name, date of on-set. Long complications are included: hernia, bleeding, bowel obstruction etc.
Extent of lymph node dissection | 2 weeks
  The extent of lymph node dissection in treatment of gastric cancer is considered a prognostic marker for postoperative survival and disease-free survival. Before implementation of a new surgical technique, it is imperative that this technique is non-inferior with regard to the extent of lymph node dissection. Measures will include the number of resected lymph nodes and the number of resected lymph node stations.

CONTACTS AND LOCATIONS:
Overall Officials: Michail Byachov, MD, PhD, Study Chair — Moscow Clinical Scientific Center; Roman Izrailov, MD, PhD, Study Chair — Moscow Clinical Scientific Center; Boris Pomortsev, MD, Principal Investigator — Moscow Clinical Scientific Center; Pavel Kononets, MD, PhD, Principal Investigator — Moscow Oncological Hospital 62; Andrey Ryabov, MD, PhD, Principal Investigator — P.Herzen Moscow Oncological Research Institute; Vladimir Lyadov, MD, PhD, Principal Investigator — Treatment and Rehabilitation Centre of Health Ministry of Russia; Alexey Karachun, MD, PhD, Principal Investigator — N. Petrov National Research Institute of Oncology; Victor Kashchenko, MD, PhD, Principal Investigator — Federal Medical Biology Agence №122 the name of L.Sokolov; Andrey Pavlenko, MD, PhD, Principal Investigator — Leningradsky oncological center; Michail Lando, MD, PhD, Principal Investigator — Lipetsk regional oncological center; Sergey Baydo, MD, PhD, Principal Investigator — Lisod clinic Kiev; Igor Khatkov, MD, PhD, Study Director — Moscow Clinical Scientific Center; Michail Prostov, Principal Investigator — Moscow Clinical Scientific Center; Kirill Schostka, MD, PhD, Principal Investigator — Leningradsky oncological center
Locations (9):
- Russia (8):
  - Lipetsk regional oncological center, Lipetsk
  - Moscow Clinical Scientific Center, Moscow
  - Moscow Oncology Hospital 62, Moscow
  - P.Herzen Moscow Oncological Research Institute, Moscow
  - Treatment and Rehabilitation Centre of Health Ministry of Russia, Moscow
  - Federal Medical Biology Agence №122 the name of L.Soko, Saint Petersburg
  - Leningradsky oncological center, Saint Petersburg
  - N. Petrov National Research Institute of Oncology, Saint Petersburg
- Lisod clinic, Kiev, Ukraine